CLINICAL TRIAL: NCT04753294
Title: A Prospective, Open, Non-comparative, Post-market Clinical Follow-up Investigation to Confirm the Safety and Performance of Avance Solo and Avance Solo Adapt NPWT Systems in Low to Moderate Exuding Chronic Wounds
Brief Title: Confirm Safety and Performance of Avance Solo and Avance Solo Adapt NPWT Systems
Acronym: ASOLO-CW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-598654
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-02

CONDITIONS: Venous Leg Ulcer; Pressure Ulcer; Diabetic Foot Ulcer; Chronic Ulcer
Keywords: Negative Pressure Wound Therapy; Post Market Clinical Follow-up
MeSH Terms: conditions — Varicose Ulcer; Pressure Ulcer; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Four different patient groups treated with the Avance Solo NPWT System or Avance Solo Adapt NPWT System.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avance Solo NPWT System (Experimental): Treatment with negative pressure wound therapy for Venous leg ulcers, Diabetic foot ulcers, and Pressure ulcers.
  Interventions: Device: Avance Solo NPWT System
- Avance Solo Adapt NPWT System (Experimental): Treatment with negative pressure wound therapy for Pressure ulcers.
  Interventions: Device: Avance Solo Adapt NPWT System

INTERVENTIONS:
Device: Avance Solo NPWT System — Wound treatment with Avance Solo NPWT System for up to 28 days.
  Arms: Avance Solo NPWT System
Device: Avance Solo Adapt NPWT System — Wound treatment with Avance Solo Adapt NPWT System for up to 28 days.
  Arms: Avance Solo Adapt NPWT System

SUMMARY:
The primary objective of this post market clinical follow-up (PMCF) investigation is to confirm the safety and performance of Avance®Solo and Avance®Solo Adapt NPWT Systems in low to moderate exuding chronic wounds when used in accordance with the Instructions for Use, for up to 28 days.

DETAILED DESCRIPTION:
This investigation is designed as a prospective, open and non-comparative PMCF investigation to confirm the safety and performance of Avance®Solo and Avance®Solo Adapt in low to moderate exuding chronic wounds. This is a multi-center study that will take place in approximately 5 European countries. The target subjects are male or female, 18 years or older with low to moderate exuding chronic wounds (pressure ulcers (N=68), diabetic foot ulcers (N=34), and venous leg ulcers (N=34)) suitable for NPWT as deemed by the investigator. Two different options of Negative Pressure Wound Therapies (NPWT) will be evaluated through this clinical investigation

A total of 136 subjects will receive treatment with the investigational devices within the intended use according to Instructions for Use (IfU): Group 1: 102 subjects in total, 34 subjects per indication (pressure ulcers, diabetic foot ulcers, and venous leg ulcers) treated with Avance®Solo and Group 2: 34 subjects with pressure ulcers treated with Avance®Solo Adapt. Subjects will be managed and monitored for a maximum of 4 weeks or until withdrawal from investigation for any reason.

The primary performance endpoint will include assessment of wound progress compared to last visit during a maximum 28 days investigation period. Wound progression is determined by the Investigator and will take into account all aspects of wound characteristics. Wound progression will be assessed by the Investigator at each follow-up visit and measured by three outcomes:

* Deteriorated
* No change
* Improved

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years.
2. Signed written informed consent.
3. Low to moderate exuding chronic wounds (diabetic foot ulcers, venous leg ulcers and pressure ulcers for Avance®Solo or pressure ulcers for Avance®Solo Adapt) suitable for NPWT according to the investigator´s judgement and Instructions for Use.
4. Subjects that will be capable and willing to comply with protocol instructions

Exclusion Criteria:

1. Known malignancy in the wound or margins of the wound
2. Untreated and previously confirmed osteomyelitis
3. Non-enteric and unexplored fistulas
4. Necrotic tissue with eschar present
5. Exposed nerves, arteries, veins or organs
6. Exposed anastomotic site
7. Known allergy/hypersensitivity to the dressing or its components.
8. Known pregnancy or planning to become pregnant or lactation at time of study participation.
9. Participation in another investigative drug or device trial currently or within the last 30 days Subjects not suitable for the investigation according to the Investigator's judgement, Clinical Investigation Plan and Instructions for Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Change in wound progress | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Wound progress compared to last visit and assessed as:
  * Deteriorated
  * No change
  * Improved

SECONDARY OUTCOMES:
Wound progress | 28 days
  Wound progress compared between baseline and final visit and assessed as:
  * Deteriorated
  * No change
  * Improved
Absolute change in wound area | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Absolute change in wound area from baseline to all follow-up visits
Absolute change in wound volume | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Absolute change in wound volume from baseline to all follow-up visits
Percentage change in wound area | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Percentage change in wound area from baseline to all follow-up visits
Percentage change in wound volume | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Percentage change in wound volume from baseline to all follow-up visits
Tissue type | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in tissue type (slough, necrotic, granulation or epithelization) from baseline to all follow-up visits.
Exudate amount | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in exudate amount using a category scoring system from baseline to all follow-up visits.
  Amount: none, low, moderate, or high)
Exudate nature | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in exudate nature using a category scoring system from baseline to all follow-up visits.
  Nature: serous, fibrinous, serosanguineous, sanguineous, seropurulent, purulent, foul purulent, heamopurulent, or hemorrhagic
Exudate odor | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in exudate odor using a category scoring system from baseline to all follow-up visits.
  Odor: no odor, slight, moderate, strong, and very strong
Peri-wound | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Change in peri-wound skin condition from baseline to all follow-up visits using the following conditions:
  * Normal
  * Erythematous
  * Oedematous
  * Eczematous
  * Excoriated
  * Macerated
  * Indurated
Tissue in-growth | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days) with additional assessments in between when dressing is changed
  Degree of tissue in-growth when Avance Solo foam is utilized at all follow-up visits as well as extra visits.
Pain assessment | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Subject evaluation of pain at Avance Solo dressing or Avance Solo Adapt Film removal using Numeric Rating Scale (NRS) at each follow-up visit.
Trauma | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Proportion of subjects with trauma to the wound site and surrounding skin for Avance Solo Border Dressing, fixation strips or Avance Solo Adapt Film at all follow-up visits.
Quality of life assessed using Numeric Rating Scale (NRS) | 28 days
  Impact of everyday life by the systems will be captured through a NRS scale where the subject grade how much the treatment has affected the subject's daily life. 0 is equal to no influence and 10 to considerable influence on everyday life or unbearable.
  If replying >0, the subject will state the presence or absence of the following causes:
  * Leakage of dressing
  * Impaired mobility
  * Difficulties in getting dressed
  * Pain
  * Odor
Alarms | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Subject evaluation of the system properties (number of sounding alarms) assessed with a given scale at all follow-up visits
  * 0
  * 1-5
  * 6-10
  * 11-15
  * 16-20
  * More than 20
Compliance | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Evaluate the compliance to the provided therapy by average number of hours per 24h that the system has not provided treatment since last visit.
Ability to absorb and/or transport exudate via clinical judgement | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Evaluation of the Systems ability to absorb and/or transport exudate assessed using a rating scale by the clinician/designee:
  * Very Poor
  * Poor
  * Good
  * Very Good
Ease of application | Baseline, Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Clinician evaluation of ease of application and removal of Avance®Solo or Avance®Solo Adapt using a Numeric Rating Scale (NRS) collected at baseline, and each follow-up visit.
Global satisfaction | 28 days
  Evaluate the investigator and subject global satisfaction of the systems in regards to:
  * Very dissatisfied
  * Dissatisfied
  * Neither satisfied or dissatisfied
  * Satisfied
  * Very satisfied
Product consumption | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Product consumption of the utilized products for the system's, from baseline and final visit using the Avance Solo or Avance Solo Adapt NPWT System
Wear time | Day 7 (+0/-2 days), Day 14 (+0/-2 days), Day 21 (+0/-2 days), and Day 28 (+0/-2 days)
  Evaluate Avance®Solo or Avance®Solo Adapt wear time in days from baseline to all follow-up visits including potential extra visits

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Beele, Prof. Dr., Principal Investigator — University Hospital, Ghent
Locations (13):
- Belgium (2):
  - Diensthoofd wondkliniek, UZ Gent, Ghent
  - AZ Delta, Roeselare
- North Zeeland Hospital, Hillerød, Denmark
- CHU Montpellier, Montpellier, France
- Germany (3):
  - Franziskus-Krankenhaus Berlin, Berlin
  - Klinik fur Dermatologie, Venerologie und Allergologie Campus Benjamin Franklin, Berlin
  - Klinikum der Ruhr-Universität Bochum, Bochum
- St James's Hospital, Dublin, Ireland
- Italy (2):
  - Ospedale San Raffaele S.r.I., Milan
  - A.O.U. Citta della Salute e della Scienza di Torino - A.O.U. Molinette San Giovanni Battista, Torino
- Portugal (3):
  - Santa casa da Misericórdia de Aveiro, Aveiro
  - Unidade de Cuidados Continuados António Francisco Guimarães, Guimarães
  - Trofa Saúde Hospital Central Hospital da Trofa, Touguinho

IPD SHARING:
Plan to Share IPD: No